CLINICAL TRIAL: NCT03476629
Title: Effects of Combined Training Versus Aerobic Training Versus Respiratory Muscle Training in Patients With Pulmonary Hypertension: A Randomized, Controlled Clinical Trial.
Brief Title: Effects of Different Types of Physical Training in Patients With Pulmonary Arterial Hypertension.
Acronym: PAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: University of Miami (Other); Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Principal Investigator, LUCIANA MARIA MALOSA SAMPAIO, Professor of the Postgraduate Program in Rehabilitation Sciences, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAH Rehabilitation
Record Dates: First submitted 2018-02-28; First posted 2018-03-26 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Arterial Hypertension; Cardiovascular Diseases; Respiratory Disease; Hypertension, Pulmonary; Pulmonary Hypertension
Keywords: Cardiopulmonary Exercise Test; Rehabilitation; Distance Traveled; Functional Capacity; Autonomic Nervous System
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Cardiovascular Diseases; Respiration Disorders; Hypertension, Pulmonary | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined Training (Experimental): Combined Training with 2 types of physical activity
  Interventions: Other: Physical activity
- Standard Training (Experimental): Physical activity with aerobic exercise
  Interventions: Other: Physical activity
- Respiratory Muscle Training (Experimental): Respiratory muscle performance
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Effects of different physical activity programs

SUMMARY:
Although there has been some progress in pharmacological management of PAH, limited functional capacity and low survival still persist, but there is evidence that exercise training can be accomplished without adverse effects or damage to cardiac function and pulmonary hemodynamics. Specifically, improvements in symptoms, exercise capacity, peripheral muscle function and quality of life. Training programs need to be better studied and well defined, and their physiological effects during physical training and functional capacity.

The aim of this study is to compare the effects of different training exercises on physical performance indicators.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is characterized by pathological changes in the pulmonary vasculature which cause an increase in pulmonary vascular resistance (PVR), restricting the flow of blood through the pulmonary circulation. It is a serious illness, progressive and usually fatal which causes significant functional limitation, mainly due to dyspnea. In order to maintain the flow of blood, pulmonary artery pressure (PAP) increases and the disease progresses leading to right ventricular dysfunction and right heart failure.

Regardless of the cause of PAH, the pulmonary arteries and arterioles have reduced capacity, and increases in cardiac output during exercise is limited. As a result, the delivery of oxygen to peripheral muscles is impaired, contributing to the symptoms of fatigue and dyspnea. While the limitation of the cardiac output to meet peripheral oxygen demand during exercise largely reduces exercise capacity, musculoskeletal dysfunction may also be involved in the exercise limitation in patients with PAH. Changes such as, muscle atrophy, decreased oxidative enzymes and a greater number of type II muscle fibers lead to an early lactic acidosis and decreased functional capacity. A modest evidence exists that exercise training can be done without adverse effects or damage to cardiac and / or pulmonary hemodynamics however, the effectiveness PAH requires more research.

ELIGIBILITY:
Inclusion Criteria:

* Having confirmed diagnosis of PAH, based on elevated pressure in the pulmonary artery measured by catheterization of the heart at rest, with WHO functional (World Health Organization's - Functional Assessment for Pulmonary Hypertension - modified after New York Heart Association Functional Classification (NYHA) functional classification) classes I, II, III or IV to capture PAH patients with pré-capillary involvement;
* Clinically stable with no previous hospitalizations in the last four weeks;
* Receiving PAH specific drug therapy for at least 3 months before the study began.

Exclusion Criteria:

* Use of continuous oxygen therapy;
* Significant musculoskeletal disease or pain / claudication members;
* Neurologic or cognitive impairment, psychiatric disorders or psychological mood (making it difficult for patients to understand the required tests);
* History of moderate or severe chronic lung disease;
* PAH patients with post-capillary involvement.
* Cardiac disease associated with cardiac failure, angina and / or unstable heart rhythm.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity | Change from Baseline to 15 weeks
  Oxygen consumption measurement during cardiopulmonary test
6 Minute Walking Test | Change from Baseline to 15 weeks
  Distance in meters
Incremental shuttle walking test | Change from Baseline to 15 weeks
  Distance in meters

SECONDARY OUTCOMES:
Autonomic Nervous System | Change from Baseline to 15 weeks
  Assesment by Heat Rate Variability analysis
Respiratory Muscle Strength | Change from Baseline to 15 weeks
  Assesment by Test of Incremental Respiratory Endurance
Musculoskeletal Function | Change from Baseline to 15 weeks
  Assesment by peripheral muscular strength testing.
Change of laboratory parameters, metabolic profile assessment and systemic inflammatory. | Change from Baseline to 15 weeks
  IL-1beta, IL-1ra, IL-6, IL-8, IL-10 and TNF-alfa (pg/ml)
Exhaled Nitric Oxide | Change from Baseline to 15 weeks
  The fraction of eNO (exhaled nitric oxide) in air will be measured by chemiluminescence
Lung function (physiological parameter) | Change from Baseline to 15 weeks
  Forced vital capacity and liters in 1 second, Total lung capacity, diffusion of carbon dioxide
Physical Activity Questionnaire (IPAQ) | Change from Baseline to 15 weeks
  The level of physical activity will be assessed using the international questionnaire short-version physical activity (IPAQ). The continuous score allows assessing energy expenditure expressed in MET minutes/week. The IPAQ categorical classifies include: Insufficiently active (does not perform any physical activity); Sufficiently active (conducts vigorous activity at least three days a week >600 MET - 1400 MET); Very active (performs more than three days per week of vigorous activity 1500 MET - 3000 MET)
Endothelial function | Change from Baseline to 15 weeks
  Endothelial function will be assessed by flow-mediated dilation (FMD)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Malosá Sampaio, Professor, Principal Investigator — University of Nove de Julho
Locations (1):
- Santa Casa de São Paulo Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Desai SA, Channick RN. Exercise in patients with pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2008 Jan-Feb;28(1):12-6. doi: 10.1097/01.HCR.0000311502.57022.73. PMID 18277824
- [Background] Schannwell CM, Steiner S, Strauer BE. Diagnostics in pulmonary hypertension. J Physiol Pharmacol. 2007 Nov;58 Suppl 5(Pt 2):591-602. PMID 18204173
- [Background] Gabbay E, Reed A, Williams TJ. Assessment and treatment of pulmonary arterial hypertension: an Australian perspective in 2006. Intern Med J. 2007 Jan;37(1):38-48. doi: 10.1111/j.1445-5994.2006.01242.x. PMID 17199843
- [Background] Rubin LJ. Primary pulmonary hypertension. N Engl J Med. 1997 Jan 9;336(2):111-7. doi: 10.1056/NEJM199701093360207. No abstract available. PMID 8988890
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M; ESC Scientific Document Group. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Heart J. 2016 Jan 1;37(1):67-119. doi: 10.1093/eurheartj/ehv317. Epub 2015 Aug 29. No abstract available. PMID 26320113
- [Background] Arena R, Lavie CJ, Milani RV, Myers J, Guazzi M. Cardiopulmonary exercise testing in patients with pulmonary arterial hypertension: an evidence-based review. J Heart Lung Transplant. 2010 Feb;29(2):159-73. doi: 10.1016/j.healun.2009.09.003. Epub 2009 Dec 6. PMID 19969471
- [Background] Naeije R. Breathing more with weaker respiratory muscles in pulmonary arterial hypertension. Eur Respir J. 2005 Jan;25(1):6-8. doi: 10.1183/09031936.04.00121004. No abstract available. PMID 15640315
- [Background] Bauer R, Dehnert C, Schoene P, Filusch A, Bartsch P, Borst MM, Katus HA, Meyer FJ. Skeletal muscle dysfunction in patients with idiopathic pulmonary arterial hypertension. Respir Med. 2007 Nov;101(11):2366-9. doi: 10.1016/j.rmed.2007.06.014. Epub 2007 Aug 6. PMID 17689235
- [Background] Mainguy V, Maltais F, Saey D, Gagnon P, Martel S, Simon M, Provencher S. Effects of a rehabilitation program on skeletal muscle function in idiopathic pulmonary arterial hypertension. J Cardiopulm Rehabil Prev. 2010 Sep-Oct;30(5):319-23. doi: 10.1097/HCR.0b013e3181d6f962. PMID 20410828
- [Background] de Man FS, Handoko ML, Groepenhoff H, van 't Hul AJ, Abbink J, Koppers RJ, Grotjohan HP, Twisk JW, Bogaard HJ, Boonstra A, Postmus PE, Westerhof N, van der Laarse WJ, Vonk-Noordegraaf A. Effects of exercise training in patients with idiopathic pulmonary arterial hypertension. Eur Respir J. 2009 Sep;34(3):669-75. doi: 10.1183/09031936.00027909. PMID 19720810
- [Background] Meyer FJ, Lossnitzer D, Kristen AV, Schoene AM, Kubler W, Katus HA, Borst MM. Respiratory muscle dysfunction in idiopathic pulmonary arterial hypertension. Eur Respir J. 2005 Jan;25(1):125-30. doi: 10.1183/09031936.04.00095804. PMID 15640333
- [Background] Kabitz HJ, Schwoerer A, Bremer HC, Sonntag F, Walterspacher S, Walker D, Schaefer V, Ehlken N, Staehler G, Halank M, Klose H, Ghofrani HA, Hoeper MM, Gruenig E, Windisch W. Impairment of respiratory muscle function in pulmonary hypertension. Clin Sci (Lond). 2008 Jan;114(2):165-71. doi: 10.1042/CS20070238. PMID 17764445
- [Background] Velez-Roa S, Ciarka A, Najem B, Vachiery JL, Naeije R, van de Borne P. Increased sympathetic nerve activity in pulmonary artery hypertension. Circulation. 2004 Sep 7;110(10):1308-12. doi: 10.1161/01.CIR.0000140724.90898.D3. Epub 2004 Aug 30. PMID 15337703
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941